CLINICAL TRIAL: NCT01705769
Title: To Evaluate the Impact of Three Feeding Regimens on the Recovery of Children From Uncomplicated Severe Acute Malnutrition (SAM) in India and to Use the Evidence to Inform National Policy
Brief Title: Effects of Three Feeding Regimens on Recovery of Uncomplicated Severely Acute Malnourished Children
Acronym: SAMPOORNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: Arth (Other); Christian Medical College, Vellore, India (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, NBhandari, Director, Society for Applied Studies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RPC538; CTRI/2012/10/003054 (Registry Identifier: Clinical Trial Registry - India)
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Uncomplicated Severe Acute Malnutrition
Keywords: treatment; severe acute malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RUTF-Centrally produced (Experimental): Ready to Use Therapeutic Food-Centrally produced by an Indian company
  Interventions: Other: Ready to Use Therapeutic Food-Centrally produced
- RUTF-Locally produced (Experimental): Ready to Use Therapeutic Food-Locally produced by the study team at each study site
  Interventions: Other: Ready to Use Therapeutic Food-Locally produced
- High energy and micronutrient rich foods (Active Comparator): High energy and micronutrient rich foods prepared by caregivers at home using ingredients provided to them
  Interventions: Other: High energy and micronutrient rich foods

INTERVENTIONS:
Other: Ready to Use Therapeutic Food-Centrally produced — Ready to Use Therapeutic Food-Centrally produced by an Indian company.
  Arms: RUTF-Centrally produced
Other: Ready to Use Therapeutic Food-Locally produced — Ready to Use Therapeutic Food prepared by the study team
  Arms: RUTF-Locally produced
Other: High energy and micronutrient rich foods — High energy and micronutrient rich foods prepared by caregivers at home using ingredients provided to them
  Arms: High energy and micronutrient rich foods

SUMMARY:
This project aims to assess the efficacy of three options under consideration in India for home management of Severe Acute Malnutrition (SAM). The investigators propose to conduct a multi-center randomized controlled trial to determine the efficacy of two community-supported home-based regimes using centrally or locally produced Ready to Use Therapeutic Foods (RUTF) for recovery from uncomplicated SAM after 16 weeks of management, compared with an augmented home-prepared foods regimen. The trial will enroll 911 children with uncomplicated SAM and will have enough statistical power to detect a 15% or greater difference in recovery rates between either one of the intervention groups compared with comparison group.

DETAILED DESCRIPTION:
India accounts for over half the global burden of severe acute malnutrition (SAM) in the world. While it is important to accelerate efforts to prevent SAM, effective management of children suffering from it is critical for reducing child mortality and achieving MDG1 and MDG4.

Available evidence mostly from studies in Africa suggest that home based management of uncomplicated SAM with Ready to Use Therapeutic Foods (RUTF) is at least as efficacious as facility-based management and that locally produced RUTF is as efficacious as centrally produced RUTF. More evidence on efficacy and effectiveness of home based management using RUTF is needed to decide if this intervention offers substantial advantages over home-prepared foods in the Indian settings. Additionally, there is a demand to generate evidence of efficacy of locally produced RUTF as compared to that of centrally produced RUTF. These issues can only be resolved through a well designed randomized controlled trial.

This project therefore aims to assess the efficacy of three options under consideration in India for home management of SAM. The investigators propose to conduct a multi-center randomized controlled trial to determine the efficacy of two community-supported home-based regimes using centrally or locally produced Ready to Use Therapeutic Foods (RUTF) for recovery from uncomplicated SAM after 16 weeks of management, compared with an augmented home-prepared foods regimen. The trial will enroll 911 children with uncomplicated SAM and will have enough statistical power to detect a 15% or greater difference in recovery rates between either one of the intervention groups compared with the comparison group.

Participants: The study will be conducted in three sites - urban slums and resettlement colonies in the national capital region, rural (predominantly tribal) Rajasthan, rural and urban Tamil Nadu. Field workers will survey the study area to measure mid-upper arm circumference (MUAC) in children 6 to 59 months of age and refer children with MUAC less than 13 cm to a study clinic. At the study clinic, anthropometric measurements will be taken and children with weight for height less than -3 SD of the WHO standards or oedema of both feet will be offered participation in the study.

Intervention and Comparison Regimes for Home Management of SAM

* Children randomized to the first intervention arm (Arm 1) will receive a centrally produced RUTF.
* Children randomized to the second intervention arm (Arm 2) will receive a locally produced RUTF.
* Children randomized to the comparison group (Arm 3) will receive augmented Home-Prepared Foods.

The amount of food advised for each child in all the 3 study arms are calculated to provide 175cal/kg body weight per day. These foods will be given to children from the time of enrollment until recovery (but not beyond 16 weeks). Caregivers of all enrolled children will receive counseling on frequency of feeding, amounts to be fed, encouraging children to continue breastfeeding and good hygiene practices. Additional support through a volunteer from the community will be provided to mothers who give consent, to assist in feeding the child.

Management Phases: The management will be in two phases:

Treatment Phase: From enrolment until recovery or 16 weeks (whichever is earlier), enrolled children will be provided the foods according to the study group they are randomized to, and counselled on their use.

Sustenance Phase: After completion of the treatment phase, children in all arms will be referred to the closest Anganwadi centre from where he/she will access supplementary foods given to children as a part of the ICDS strategy. The sustenance phase will last for 16 weeks after end of treatment phase.

Outcomes: A trained and standardized team of field workers will conduct weekly anthropometric measurements and also record morbidity, hospitalizations and deaths from enrolment, weekly till recovery or 16 weeks whichever is earlier. In addition, mortality and hospitalization data will be collected at 16 weeks post treatment phase.

The primary outcome will be recovery by 16 weeks after enrollment (defined as achieving weight for height greater than or equal to -2 SD and absence of oedema).

Secondary outcomes will include:

* To compare the weight gain (in grams/kg body weight/day) from enrolment till recovery, or till 16 weeks in those who do not attain recovery, at 16 weeks after recovery.
* To compare the time required to reach recovery (in weeks).
* To determine the incidence and prevalence of diarrhea, ARI and fever during the treatment phase
* To compare the mortality and hospitalizations during the treatment phase, 16 weeks after recovery
* To compare the perceptions of families, health care providers and ICDS functionaries regarding feasibility of use of the feeding regimens in a sub sample from enrolment tom completion of treatment phase
* To ascertain factors which affect recovery, at 16 weeks post enrolment in those who do not recover.
* To compare the perceptions of families regarding Anganwadi centre experience at the end of sustenance phase.
* To compare the proportion of children with weight for height greater than or equal to -2 SD and absence of oedema feet at 16 weeks after recovery (or 32 weeks after enrolment for those who do not recover)
* To document the costs of implementing the feeding regimens till end of treatment phase.

This will include:

1. Estimation of costs of human resource and other inputs
2. Estimation of household costs
3. Costs per week per child estimated based on total costs and covered population

The project has been approved by the National Research Alliance for SAM constituted by the Department of Health and Family Welfare, Department of Health Research and Department of Biotechnology. It will be coordinated by Centre for Health Research and Development-Society for Applied Studies. WHO will provide technical support and monitoring for the study implementation as a response to a request from the Alliance. Oversight to the study will be provided by a Technical Advisory group constituted by the Alliance and a Data Safety Monitoring Board. Clearances have been sought from the state governments of Delhi, Rajasthan and Tamil Nadu.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 59 months
* SAM, defined as Weight for height less than -3 SD of WHO standard or oedema of both feet or both.

Exclusion Criteria:

* Complicated SAM defined as child with SAM having signs of severe illness requiring hospitalization
* Known allergy to animal milk or peanuts
* Likely to leave the study area permanently in the next 16 weeks

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 911 (Actual)
Dates: Start 2012-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Recovery by 16 weeks after enrollment (defined as achieving weight for height greater than or equal to -2 SD and absence of oedema of both feet) | Weekly till recovery or 16 weeks after enrollment, whichever is earlier

SECONDARY OUTCOMES:
Mortality and hospitalizations | Weekly till 16 weeks or recovery and at end of sustenance phase
Rate of weight gain (grams/kg body wt/day) | From enrollment till recovery or 16 weeks whichever is earlier
Time required to reach recovery | From enrollment till recovery or 16 weeks whichever is earlier
Íncidence and prevalence of diarrhea, ARI and fever during treatment phase | From enrollment till recovery or 16 weeks whichever is earlier
Proportion of children with weight for height greater than or equal to -2 SD and absence of oedema of feet | At the end of sustenance phase
Cost of three feeding regimens | Enrollment to end of treatment phase
Feedback from families, health care providers and ICDS functionaries about the feeding regimens regarding perceptions and feasibility of use | Enrollment to end study
Factors which affect recovery | At 16 weeks post enrolment in those that have not recovered
Perception of families regarding anganwadi centre experiences at the end of sustenance phase | from end of treatment phase to end of sustanence phase

CONTACTS AND LOCATIONS:
Overall Officials: Nita Bhandari, MD, PhD, Principal Investigator — Centre for Health Research and Development, Society for Applied Studies
Locations (3):
- India (3):
  - Centre for Health Research and Development, Society for Applied Studies, New Delhi, National Capital Territory of Delhi
  - Action Research & Training for Health (ARTH), Udaipur, Rajasthan
  - Christian Medical College, Vellore, Tamil Nadu

REFERENCES:
- [Derived] Garg CC, Mazumder S, Taneja S, Shekhar M, Mohan SB, Bose A, Iyengar SD, Bahl R, Martines J, Bhandari N. Costing of three feeding regimens for home-based management of children with uncomplicated severe acute malnutrition from a randomised trial in India. BMJ Glob Health. 2018 Mar 6;3(2):e000702. doi: 10.1136/bmjgh-2017-000702. eCollection 2018. PMID 29527358
- [Derived] Bhandari N, Mohan SB, Bose A, Iyengar SD, Taneja S, Mazumder S, Pricilla RA, Iyengar K, Sachdev HS, Mohan VR, Suhalka V, Yoshida S, Martines J, Bahl R. Efficacy of three feeding regimens for home-based management of children with uncomplicated severe acute malnutrition: a randomised trial in India. BMJ Glob Health. 2016 Dec 30;1(4):e000144. doi: 10.1136/bmjgh-2016-000144. eCollection 2016. PMID 28588982